CLINICAL TRIAL: NCT05216406
Title: Effects of Daily Supplementation of 5-HTP on Body Composition, a Randomized Investigation
Brief Title: Effects of Daily Supplementation of 5-HTP on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Cassandra Evans, Co-principal Investigator, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 102
Record Dates: First submitted 2021-12-07; First posted 2022-01-31 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Body Composition
Keywords: Body Composition; 5-HTP
MeSH Terms: interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Intervention Model Description: This study followed a placebo (PLA)-controlled, double-blind and parallel-group design.
Who Masked: Participant, Investigator
Masking Description: All subjects and investigators were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-HTP (Experimental): The dietary supplement (100 mg of 5-hydroxytryptophan; CLEANMOOD™) was provided by NURA™ (Irvine, California USA). Subjects were instructed to consume one capsule daily at their convenience for 8 weeks.
  Interventions: Dietary Supplement: 5-HTP
- Control (Placebo Comparator): The placebo consisted of maltodextrin. Subjects were instructed to consume one capsule daily at their convenience for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 5-HTP — CLEANMOOD is an organic 5-Hydroxytryptophan (5-HTP) ingredient.
  Other Names: CLEANMOOD™
  Arms: 5-HTP
Other: Placebo — Maltodextrin capsule
  Other Names: Control
  Arms: Control

SUMMARY:
The purpose of this investigation was to compare supplementation with 5-HTP to placebo on indices of body composition. A randomized trial compared a sample of 48 resistance-trained individuals taking either 100 mg of 5-hydroxytryptophan supplementation or a placebo.

The investigators tested anthropometric measurements using a multi-frequency bioelectrical impedance device (InBody® 270). The primary outcome (i.e., changes in anthropometric measurements) was assessed at the first visit (pre-test-) and post-test (8 weeks). Secondary outcomes include resting heart rate, blood pressure, and dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or free of disease
* Minimum of 1 year of regular physical activity. Regular physical activity is defined by a minimum of 150 minutes of aerobic activity or performing muscle-strengthening exercises at least 2 days a week.

Exclusion Criteria:

* Physically inactive
* Regularly used sleep aids of any kind
* Currently taking selective serotonin reuptake inhibitors (SSRIs) and/or 5-HTP containing supplements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- IHP, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maffei ME. 5-Hydroxytryptophan (5-HTP): Natural Occurrence, Analysis, Biosynthesis, Biotechnology, Physiology and Toxicology. Int J Mol Sci. 2020 Dec 26;22(1):181. doi: 10.3390/ijms22010181. PMID 33375373
- [Background] Stamatakis E, Straker L, Hamer M, Gebel K. The 2018 Physical Activity Guidelines for Americans: What's New? Implications for Clinicians and the Public. J Orthop Sports Phys Ther. 2019 Jul;49(7):487-490. doi: 10.2519/jospt.2019.0609. PMID 31258047
- [Background] Cangiano C, Ceci F, Cairella M, Cascino A, Del Ben M, Laviano A, Muscaritoli M, Rossi-Fanelli F. Effects of 5-hydroxytryptophan on eating behavior and adherence to dietary prescriptions in obese adult subjects. Adv Exp Med Biol. 1991;294:591-3. doi: 10.1007/978-1-4684-5952-4_73. No abstract available. PMID 1722953

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5-HTP | Control
Started | 39 | 26
Completed | 31 | 17
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-HTP | Control | Total
Number analyzed (Participants) | 31 | 17 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 17 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 12 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Composition [Mean (Standard Deviation); unit: Kilograms]
  Fat Mass | 15.3 (6.0) | 12.4 (4.4) | 13.9 (5.2)
  Lean Body Mass | 57.5 (13.9) | 57.5 (13.7) | 57.5 (13.8)
  Body Mass | 72.9 (13.4) | 69.1 (11.9) | 71 (12)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 118 (14) | 117 (13) | 117.5 (13.5)
  Diastolic | 72 (10) | 70 (6) | 71 (4)
Resting Heart Rate [Mean (Standard Deviation); unit: Beats Per Minute (BPM)] | 69 (12) | 70 (13) | 69.5 (10)
Dietary Intake [Mean (Standard Deviation); unit: Kilocalories]
  Total Intake | 1906 (683) | 2022 (765) | 1964 (720)
  Fat | 603 (288) | 630 (234) | 616.5 (261)
  Carbohydrate | 836 (452) | 840 (424) | 838 (438)
  Protein | 468 (172) | 548 (224) | 508 (198)

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: The percentage of fat, bone, and muscle was assessed pre and post visit using multi-frequency bioelectrical impedance device (InBody® 270).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | 5-HTP | Control
Number analyzed (Participants) | 31 | 17
Kilograms
  Fat Mass | 14.6 (5.7) | 12.6 (4.4)
  Lean Body Mass | 58.4 (13.9) | 57.7 (13.6)
  Body Mass | 73 (12.8) | 70.2 (12.4)

2. Secondary Outcome: Dietary Habits
Description: The mobile app MyFitnessPal was used to assess dietary intake. Subjects were instructed to log their food intake MyFitnessPal, for a minimum of 2-3 days per week during the entire study.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | 5-HTP | Control
Number analyzed (Participants) | 31 | 17
calories
  Total Intake | 1810 (650) | 1966 (826)
  Fat | 576 (198) | 684 (387)
  Carbohydrate | 796 (364) | 816 (392)
  Protein | 440 (140) | 464 (168)

3. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure will be measured during pre and post visit using an upper arm blood pressure monitor and cuff.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | 5-HTP | Control
Number analyzed (Participants) | 31 | 17
mmHG
  Systolic | 119 (14) | 117 (16)
  Diastolic | 70 (7) | 67 (11)

4. Secondary Outcome: Resting Heart Rate
Description: Resting heart rate will be measured pre and post visit using an upper arm blood pressure monitor and cuff.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | 5-HTP | Control
Number analyzed (Participants) | 31 | 17
BPM | 70 (10) | 65 (7)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Self-report at the end of the trial.
Arm/Group | 5-HTP | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/17
Other Adverse Events (participants affected / at risk) | 3/31 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-HTP (N=31) | Control (N=17)
Upset Stomach (Gastrointestinal disorders) | 3 (3) | 2 (2) — a disorder of digestive function characterized by discomfort or heartburn or nausea. dyspepsia, indigestion, stomach upset

LIMITATIONS AND CAVEATS:
The primary limitation of this study was the lack of control for exercise. Although subjects were instructed to maintain the same training habits, it is certainly possible that training changed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05216406/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT05216406/ICF_000.pdf